CLINICAL TRIAL: NCT05854316
Title: Protocols and Guidelines for the Use of Digital Twins in Frail Older People
Acronym: Proto-Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Proto-Aging
Record Dates: First submitted 2023-04-19; First posted 2023-05-11 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Frail Elderly Syndrome
Keywords: Elderly; Frailty; Dynapenia; Muscle weakness; Maximal Voluntary Isometric Contraction; Superimposed Neuromuscular Electrical Stimulation; Dynamometry; Electromyography; Clinical questionnaires; Hand-grip test
MeSH Terms: conditions — Frailty; Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Frail elders (Experimental): Frail elders; Age: 65-80 years; Body Mass Index: 18.5-30 kg/m²; Frailty diagnosed according to Fried's criteria (i.e., at least three of the following items: unintended loss of weight, weakness, self-reported exhaustion, slow walking speed, low level of physical activity).
  Interventions: Diagnostic Test: Comprehensive Biomechanical assessment

INTERVENTIONS:
Diagnostic Test: Comprehensive Biomechanical assessment — Magnetic resonance images, electromyography and dynamometry data will be used, together with data from the gait assessment and clinical questionnaires/measures, to characterize the biomechanics of the participants, and to develop and inform personalised musculoskeletal models

SUMMARY:
The Proto-Aging study aims to define experimental protocols and guidelines to enable the development of musculoskeletal models (digital twins) of elderly people, with the ultimate goal to comprehensively characterize frail elders from a biomechanical standpoint.

It is typical for the elderly to present with weakness, slowed movements and reduced levels of physical activity, all of which may be related to the loss of muscle force (dynapenia). Unfortunately, to date, the primary cause for dynapenia is difficult to identify. Digital twins may help to this end, but their development remains critical as it requires a specialized skillset and experimental data for model personalisation.

In this study, where the investigators will recruit a small group of frail elders and a cohort of healthy young individuals, all participants will undergo the following examinations: (i) gait assessment, (ii) maximal voluntary isometric contraction (MVIC) test, (iii) superimposed neuromuscular electrical stimulation, and (iv) full lower limb magnetic resonance imaging. Surface electromyography data will further be collected while the subjects perform both the gait assessment and the MVIC test. Last, clinical questionnaires will be administered, and the subjects will be asked to perform additional clinical measures (i.e., hand-grip test, bioelectrical impedance analysis).

At the end of the study, a reduced version of the experimental protocol will be developed, with the intent to provide clinicians with a protocol that can be deployed in clinical settings, accounting for the observed reliability and repeatability of each measure, the required level of expertise, and the associated costs and time expenditure.

ELIGIBILITY:
Inclusion Criteria:

* Age: 65-80 years
* Body Mass Index between 18.5 and 30 kg/m2
* Frailty syndrome diagnosed according to Fried's criteria (i.e., at least three of the following items: unintended loss of weight, weakness, self-reported exhaustion, slow walking speed, low level of physical activity)

Exclusion Criteria:

* Any musculoskeletal, neurological, rheumatic or tumoral diseases
* Dementia
* Diabetes
* Inguinal or abdominal hernia
* Severe Hypertension (Level 3)
* Severe Cardio-pulmonary insufficiency
* Diagnosis of Osteonecrosis in the lower limb joints
* Pathologies or physical conditions incompatible with the use of magnetic resonance imaging and electrostimulation (i.e., active and passive implanted biomedical devices, epilepsy, severe venous insufficiency in the lower limbs)
* Previous interventions or traumas to the joints of the lower limb

NOTE: A group of healthy volunteers, who meet the following criteria, will be enrolled in the study:

Inclusion Criteria:

* Age: 20-40 years;
* Body Mass Index: 15-30 kg/m²;
* Physical activity level (Saltin-Grimby): 2-4
* No previous or known musculoskeletal, neurological, rheumatic or tumoral diseases

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Muscle volume | at baseline (Day 0)
  Full lower limb MRI data will be acquired with subjects in supine position. Individual muscle volumes (in cm3) will be segmented using commercial software and stored in anonymized form.
MVIC Torque | at baseline (Day 0)
  Dynamometry data will be acquired while participants perform a MVIC leg extension test. The maximum torque values (Nm) measured over three repetitions will be recorded. These correspond to the values observed in correspondence of the plateaux of force, developed over a sustained contraction
Muscle Inhibition level | at baseline (Day 0)
  The difference between the maximal force exerted during the MVIC test (voluntary contraction) and that achieved when the muscles are electrically stimulated (involuntary contraction) will be computed
Co-contraction index (CCI) | at baseline (Day 0)
  Experimental EMG data will be recorded from the major lower limb muscles involved in the knee extension, while participants perform a maximal voluntary isometric contraction on a dynamometer (i.e., MVIC test to quantify muscle strength). The co-contraction index, defined as the relative activation of agonist and antagonist muscles (for this task: quadriceps and hamstrings) in the act of kicking (MVIC test).
Body kinematics | at baseline (Day 0)
  A standard gait assessment will be performed where motion capture data will be collected. Joint angles will be extracted to identify abnormal gait patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Benedetti, Professor, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy